CLINICAL TRIAL: NCT05827614
Title: An Open-Label, Multicenter, First-in-Human, Dose-Escalation and Dose-Expansion, Phase 1/2 Study of BBI-355 and BBI-355 in Combination With Select Targeted Therapies in Subjects With Locally Advanced or Metastatic Solid Tumors With Oncogene Amplifications
Brief Title: Study of the CHK1 Inhibitor BBI-355, an ecDNA-directed Therapy (ecDTx), and the RNR Inhibitor BBI-825, in Subjects With Tumors With Oncogene Amplifications
Acronym: POTENTIATE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boundless Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BBI-355-101
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer (TNBC); High Grade Serous Ovarian Carcinoma; High Grade Endometrial Carcinoma; Anogenital Cancer; Head and Neck (HNSCC); Cutaneous Squamous Cell Carcinoma (CSCC); Cervical Squamous Cell Carcinoma; ER+ Breast Cancer; Leiomyosarcoma (LMS); Undifferentiated Pleomorphic Sarcoma (UPS); Pancreatic Cancer Metastatic; Small Cell Lung Cancer
Keywords: ecDNA; extrachromosomal DNA; Amplification; Oncogene Amplification; Checkpoint kinase 1; CHK1; RNR; ribonucleotide reductase
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Leiomyosarcoma; Histiocytoma, Malignant Fibrous; Small Cell Lung Carcinoma | interventions — Erlotinib Hydrochloride; futibatinib

STUDY DESIGN:
Intervention Model Description: BBI-355 single agent dose escalation and expansion, and BBI-355 dose escalation in combination with select targeted therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single Agent Dose Escalation (Experimental): Single agent BBI-355, administered orally in 28-day cycles
  Interventions: Drug: BBI-355
- Single Agent Dose Expansion (Experimental): Single agent BBI-355, administered orally in 28-day cycles
  Interventions: Drug: BBI-355
- Dose Escalation in Combination with EGFR Inhibitor (Experimental): Combination therapy of BBI-355 and EGFR inhibitor erlotinib, administered orally in 28-day cycles.
  Interventions: Drug: BBI-355; Drug: Erlotinib
- Dose Escalation in Combination with FGFR Inhibitor (Experimental): Combination therapy of BBI-355 and FGFR1-4 inhibitor futibatinib, administered orally in 28-day cycles.
  Interventions: Drug: BBI-355; Drug: Futibatinib
- Dose Escalation in Combination with RNR Inhibitor (Experimental): Combination therapy of BBI-355 and RNR Inhibitor BBI-825, administered orally in 28-day cycles.
  Interventions: Drug: BBI-355; Drug: BBI-825

INTERVENTIONS:
Drug: BBI-355 — Oral CHK1 inhibitor
Drug: Erlotinib — EGFR Inhibitor
  Arms: Dose Escalation in Combination with EGFR Inhibitor
Drug: Futibatinib — FGFR1-4 Inhibitor
  Arms: Dose Escalation in Combination with FGFR Inhibitor
Drug: BBI-825 — Oral RNR Inhibitor
  Arms: Dose Escalation in Combination with RNR Inhibitor

SUMMARY:
BBI-355 is an oral, potent, selective checkpoint kinase 1 (or CHK1) small molecule inhibitor in development as an ecDNA (extrachromosomal DNA) directed therapy (ecDTx). BBI-825 is an oral, potent, selective ribonucleotide reductase (or RNR) small molecule inhibitor. This is a first-in-human, open-label, 2-part, Phase 1/2 study to determine the safety profile and identify the maximum tolerated dose and recommended Phase 2 dose of BBI-355 administered as a single agent or in combination with BBI-825 or other select therapies.

DETAILED DESCRIPTION:
BBI-355 and BBI-825 are administered orally in various dosing schedules to subjects with locally advanced or metastatic non-resectable solid tumors harboring oncogene amplifications, whose disease has progressed despite all standard therapies or for whom no further standard or clinically acceptable therapy exists.

ELIGIBILITY:
Key Inclusion Criteria:

* Locally advanced or metastatic non-resectable solid tumors, whose disease has progressed despite all standard therapies or for whom no further standard or clinically acceptable therapy exists,
* Evidence of oncogene amplification,
* Availability of FFPE tumor tissue, archival or newly obtained,
* Measurable disease as defined by RECIST Version 1.1,
* Adequate hematologic function,
* Adequate hepatic and renal function,
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1,
* Other inclusion criteria per study protocol.

Key Exclusion Criteria:

* Single agent arm: Prior exposure to CHK1 or WEE1 inhibitors,
* BBI-355 combination with BBI-825 arm: Prior exposure to combination therapy of any RNR inhibitor plus CHK1/2 inhibitor,
* Hematologic malignancies,
* Primary CNS malignancy, leptomeningeal disease, or symptomatic active CNS metastases, with exceptions per study protocol,
* Prior or concurrent malignancies, with exceptions per study protocol,
* History of HBV, HCV, or HIV infection,
* Clinically significant cardiac condition,
* Active or history of interstitial lung disease (ILD) or pneumonitis, or history of ILD or pneumonitis requiring steroids or other immunosuppressive medications,
* QTcF > 470 msec,
* Prior organ allograft transplantations or allogeneic peripheral blood stem cell/bone marrow transplantation,
* Other exclusion criteria per study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs) of BBI-355 as a single agent and in combination with each of the following agents: erlotinib, futibatinib, or BBI-825 | Start of Cycle 1 until 30 days following last dose (each cycle is 28 days)
  TEAEs will be assessed and severity assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of BBI-355 as a single agent and in combination with erlotinib, futibatinib, or BBI-825 | Start of Cycle 1 until 30 days following last dose (each cycle is 28 days)
  The MTD and/or RP2D of BBI-355 as a single agent and in combination with erlotinib, futibatinib, or BBI-825 will be determined.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BBI-355, erlotinib, futibatinib, and BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Maximum observed plasma concentration (Cmax) of BBI-355, erlotinib, futibatinib, and BBI-825 will be determined.
Trough observed plasma concentration (Ctrough) of BBI-355, erlotinib, futibatinib, and BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Trough observed plasma concentration (Ctrough) of BBI-355, erlotinib, futibatinib and BBI-825 will be determined.
Time to Cmax (Tmax) of BBI-355, erlotinib, futibatinib, and BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Time to Cmax (Tmax) of BBI-355, erlotinib, futibatinib, and BBI-825 will be determined.
Area under the concentration time curve (AUC) of BBI-355, erlotinib, futibatinib, and BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Area under the concentration time curve (AUC) of BBI-355, erlotinib, futibatinib and BBI-825 will be determined.
Anti-tumor activity of BBI-355 as a single agent and in combination with erlotinib, futibatinib, or BBI-825 | 1-2 years: Start of Cycle 1 until documented disease progression or death (each cycle is 28 days)
  Tumor response will be determined by RECISTv1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Doebele, MD, PhD, Study Director — Boundless Bio
Locations (16):
- United States (16):
  - UCLA Medical Center, Los Angeles, California
  - Sarcoma Oncology, Santa Monica, California
  - HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Lake Mary, Florida
  - The University of Kansas, Fairway, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology - Dallas, Irving, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
  - University of Washington, Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones R, Plummer R, Moreno V, Carter L, Roda D, Garralda E, Kristeleit R, Sarker D, Arkenau T, Roxburgh P, Walter HS, Blagden S, Anthoney A, Klencke BJ, Kowalski MM, Banerji U. A Phase I/II Trial of Oral SRA737 (a Chk1 Inhibitor) Given in Combination with Low-Dose Gemcitabine in Patients with Advanced Cancer. Clin Cancer Res. 2023 Jan 17;29(2):331-340. doi: 10.1158/1078-0432.CCR-22-2074. PMID 36378548
- [Background] Italiano A, Infante JR, Shapiro GI, Moore KN, LoRusso PM, Hamilton E, Cousin S, Toulmonde M, Postel-Vinay S, Tolaney S, Blackwood EM, Mahrus S, Peale FV, Lu X, Moein A, Epler J, DuPree K, Tagen M, Murray ER, Schutzman JL, Lauchle JO, Hollebecque A, Soria JC. Phase I study of the checkpoint kinase 1 inhibitor GDC-0575 in combination with gemcitabine in patients with refractory solid tumors. Ann Oncol. 2018 May 1;29(5):1304-1311. doi: 10.1093/annonc/mdy076. PMID 29788155
- [Background] Tang J, Weiser NE, Wang G, Chowdhry S, Curtis EJ, Zhao Y, Wong IT, Marinov GK, Li R, Hanoian P, Tse E, Mojica SG, Hansen R, Plum J, Steffy A, Milutinovic S, Meyer ST, Luebeck J, Wang Y, Zhang S, Altemose N, Curtis C, Greenleaf WJ, Bafna V, Benkovic SJ, Pinkerton AB, Kasibhatla S, Hassig CA, Mischel PS, Chang HY. Enhancing transcription-replication conflict targets ecDNA-positive cancers. Nature. 2024 Nov;635(8037):210-218. doi: 10.1038/s41586-024-07802-5. Epub 2024 Nov 6. PMID 39506153
- [Background] Wu S, Bafna V, Chang HY, Mischel PS. Extrachromosomal DNA: An Emerging Hallmark in Human Cancer. Annu Rev Pathol. 2022 Jan 24;17:367-386. doi: 10.1146/annurev-pathmechdis-051821-114223. Epub 2021 Nov 9. PMID 34752712
- [Background] Turner KM, Deshpande V, Beyter D, Koga T, Rusert J, Lee C, Li B, Arden K, Ren B, Nathanson DA, Kornblum HI, Taylor MD, Kaushal S, Cavenee WK, Wechsler-Reya R, Furnari FB, Vandenberg SR, Rao PN, Wahl GM, Bafna V, Mischel PS. Extrachromosomal oncogene amplification drives tumour evolution and genetic heterogeneity. Nature. 2017 Mar 2;543(7643):122-125. doi: 10.1038/nature21356. Epub 2017 Feb 8. PMID 28178237
- [Background] Lange JT, Rose JC, Chen CY, Pichugin Y, Xie L, Tang J, Hung KL, Yost KE, Shi Q, Erb ML, Rajkumar U, Wu S, Taschner-Mandl S, Bernkopf M, Swanton C, Liu Z, Huang W, Chang HY, Bafna V, Henssen AG, Werner B, Mischel PS. The evolutionary dynamics of extrachromosomal DNA in human cancers. Nat Genet. 2022 Oct;54(10):1527-1533. doi: 10.1038/s41588-022-01177-x. Epub 2022 Sep 19. PMID 36123406
- [Background] Kim H, Nguyen NP, Turner K, Wu S, Gujar AD, Luebeck J, Liu J, Deshpande V, Rajkumar U, Namburi S, Amin SB, Yi E, Menghi F, Schulte JH, Henssen AG, Chang HY, Beck CR, Mischel PS, Bafna V, Verhaak RGW. Extrachromosomal DNA is associated with oncogene amplification and poor outcome across multiple cancers. Nat Genet. 2020 Sep;52(9):891-897. doi: 10.1038/s41588-020-0678-2. Epub 2020 Aug 17. PMID 32807987